CLINICAL TRIAL: NCT04947683
Title: Patient Journey With Advanced Lung Cancer Positive for ALK Fusion in Brazil
Acronym: ALK
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 1918
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma; Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, retrospective cohort study that will include patients diagnosed with NSCLC and ALK rearrangement between January 2015 and December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years;
* Newly diagnosed advanced stage IIIB-IV NSCLC (AJCC 8th edition) or locally advance/distant relapse in the period of January 2015 to December 2020.
* NSCLC with pathological confirmation of ALK rearrangement by immunohistochemistry, fluorescent in situ hybridization (FISH) or next generation sequencing (NGS);
* ECOG 0-4;
* Patients with CNS metastases are also considered eligible, regardless of the initial treatment instituted.

Exclusion Criteria:

- Incomplete medical chart in terms of date of diagnosis, ALK test results and outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic patients with NSCLC and ALK rearrangement between January 2015 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
- Describe the treatment sequencing of ALK positive advanced NSCLC in a real-world setting. | December of 2020
- Describe the timelines from the appearance of symptoms, histopathological diagnosis, application of the molecular test, and start of treatment. | December of 2020

SECONDARY OUTCOMES:
- Estimate the progression-free survival of first-line treatment, and other subsequent lines; | December of 2020

OTHER OUTCOMES:
- Estimate the overall survival from diagnosis | December of 2020
- Compare patients' outcomes among baseline characteristics defined subgroups; | December of 2020
- Evaluate health economics parameters in the context. | December of 2020

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Centro Regional Integrado de Oncologia (CRIO), Fortaleza, Ceará
  - Instituto D'OR, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - CPO Pucrs, Porto Alegre, Rio Grande do Sul
  - A.C Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: No